CLINICAL TRIAL: NCT05876923
Title: The Effects of Acute and Chronic Exercise on the Immune Phenotype of Indolent Non-Hodgkin Lymphoma and Chronic Lymphocytic Leukemia Patients
Brief Title: The Effects of Exercise on Immune Phenotype of Indolent Non-Hodgkin Lymphoma and Chronic Lymphocytic Leukemia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-012246; NCI-2023-03210 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-012246 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-05-01; First posted 2023-05-26 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma; Indolent Non-hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Specimen Handling; Exercise Test; Clostridium perfringens epsilon-toxin; Absorptiometry, Photon; Bone Density; Restraint, Physical; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Aim 1 (vitals, spirometry, CPET, blood samples, DEXA) (Experimental): Participants undergo measurement of height/weight and vital signs (blood pressure, temperature, heart and breathing rate), complete lung function testing (spirometry), undergo an exercise test (CPET), and undergo collection of blood samples on study. Participants may also undergo DEXA scan on study.
  Interventions: Procedure: Biospecimen Collection; Other: Cardiopulmonary Exercise Testing; Procedure: Dual X-ray Absorptiometry; Other: Electronic Health Record Review; Procedure: Physical Examination; Other: Questionnaire Administration; Procedure: Spirometry
- Aim 2 (aerobic based training program, Aim 1 activities) (Experimental): CLL patients complete aerobic based training program on study. Patients then complete all Aim 1 activities again after completion of aerobic based training program.
  Interventions: Procedure: Biospecimen Collection; Other: Cardiopulmonary Exercise Testing; Procedure: Dual X-ray Absorptiometry; Other: Electronic Health Record Review; Other: Exercise Intervention; Procedure: Physical Examination; Other: Questionnaire Administration; Procedure: Spirometry
- Aims 3-4 arm I (indolent NHL usual care) (Active Comparator): Indolent NHL patients undergo measurement of height/weight and vital signs (blood pressure, temperature, heart and breathing rate), complete lung function testing (spirometry), undergo an exercise test (CPET), and undergo collection of blood samples on study. Participants may also undergo DEXA scan on study. Patients undergo muscular strength and functional endurance measurements of hand grip strength, upper body power via weighted chest pass, and leg strength with the timed chair stand test and 6MWT. Patients receive usual care on study.
  Interventions: Procedure: Biospecimen Collection; Other: Cardiopulmonary Exercise Testing; Procedure: Dual X-ray Absorptiometry; Other: Electronic Health Record Review; Procedure: Physical Examination; Other: Questionnaire Administration; Procedure: Spirometry; Other: Physical Performance Testing; Other: Best Practice
- Aims 3-4 arm II (indolent NHL aerobic based training program) (Active Comparator): Indolent NHL patients undergo measurement of height/weight and vital signs (blood pressure, temperature, heart and breathing rate), complete lung function testing (spirometry), undergo an exercise test (CPET), and undergo collection of blood samples on study. Participants may also undergo DEXA scan on study. Patients undergo muscular strength and functional endurance measurements of hand grip strength, upper body power via weighted chest pass, and leg strength with the timed chair stand test and 6MWT. Patients complete aerobic based training program on study. Patients then complete all baseline activities again after completion of aerobic based training program.
  Interventions: Procedure: Biospecimen Collection; Other: Cardiopulmonary Exercise Testing; Procedure: Dual X-ray Absorptiometry; Other: Electronic Health Record Review; Other: Exercise Intervention; Procedure: Physical Examination; Other: Questionnaire Administration; Procedure: Spirometry; Other: Physical Performance Testing; Other: Best Practice
- Aim 5 (repeat baseline activities) (Experimental): All patients from Aims 3-4 will be invited to repeat Aims 3-4 baseline activities.
  Interventions: Procedure: Biospecimen Collection; Other: Cardiopulmonary Exercise Testing; Procedure: Dual X-ray Absorptiometry; Other: Electronic Health Record Review; Procedure: Physical Examination; Other: Questionnaire Administration; Procedure: Spirometry; Other: Physical Performance Testing

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Cardiopulmonary Exercise Testing — Undergo CPET
  Other Names: CPET; CPX
Procedure: Dual X-ray Absorptiometry — Undergo DEXA scan
  Other Names: BMD scan; bone mineral density scan; DEXA; DEXA (Bone Density); DEXA Scan; dual energy x-ray absorptiometric scan; Dual Energy X-ray Absorptiometry; Dual X-Ray Absorptometry; DXA; DXA SCAN
Other: Electronic Health Record Review — Ancillary studies
Other: Exercise Intervention — Undergo aerobic based training program
  Arms: Aim 2 (aerobic based training program, Aim 1 activities); Aims 3-4 arm II (indolent NHL aerobic based training program)
Procedure: Physical Examination — Undergo measurement of height/weight and vital signs
  Other Names: Assessment; General Examination; Physical; Physical Assessment; Physical Exam; Physical examination procedure (procedure); physical_exam
Other: Questionnaire Administration — Ancillary studies
Procedure: Spirometry — Undergo spirometry
Other: Physical Performance Testing — Undergo muscular strength and functional endurance measurements
  Other Names: Physical Fitness Testing; Physical Function Testing
  Arms: Aim 5 (repeat baseline activities); Aims 3-4 arm I (indolent NHL usual care); Aims 3-4 arm II (indolent NHL aerobic based training program)
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Aims 3-4 arm I (indolent NHL usual care); Aims 3-4 arm II (indolent NHL aerobic based training program)

SUMMARY:
This clinical trial studies the effect of short-term (acute) and long-term (chronic) exercise on immune characteristics and function (phenotype) of patients with indolent non-Hodgkin lymphoma (NHL) and chronic lymphocytic leukemia (CLL). Most newly-diagnosed CLL patients have early-stage disease at the time of diagnosis and do not require treatment. Despite not needing therapy, these patients have significant immune dysfunction. This may lead to an increased risk of serious infections requiring hospitalization and an increased risk of secondary non-blood-based (hematologic) cancers. Increasing CLL patients overall physical fitness levels, through exercise during the observation stage, may provide a realistic approach means to increase survival, decrease treatment-related side effects, and improve immune function. Information learned from this study may help researchers determine whether a particular exercise regimen can be used to strengthen the immune system of indolent NHL and CLL patients, delay time to disease progression, assess the need for treatment, and assess infection rates.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine how circulating immune cell abundance and function (via cell counts & cytokine profile) of CLL patients respond to acute (single bout) maximal exercise and how this differs from the response observed in group of age-matched controls by monitoring cardiopulmonary parameters and mobilization of immune cell phenotypes.

II. Determine how circulating immune cell mobilization and function (cell counts & cytokine profile) of CLL patients respond to a 12-week semi-supervised training program of moderate to high intensity, aerobic based exercise.

III. Evaluate the effectiveness of 12-weeks of semi-supervised exercise training (ET) versus (vs.) usual care (UC) at reducing cancer-related side effects and improving quality of life (QOL) and physical fitness in individuals with indolent non-Hodgkin (NHL) lymphoma during or after treatment.

IV. Determine that extent to which 12-weeks of semi-supervised ET can modify circulating immune cell mobilization and immune function in individuals with indolent NHL during or after treatment compared to UC.

V. Development of a forward-chaining AI expert system using both manual and physiology derived feedback to optimize training results and compare its efficacy at reducing cancer-related side effects and improving quality of life (QOL) and physical fitness in individuals with indolent NHL and CLL to that of the semi-supervised ET.

OUTLINE: CLL patients and healthy participants are assigned to Aim 1. CLL patients who complete all Aim 1 activities are assigned to Aim 2. Patients with indolent NHL will be assigned to Aims 3 and 4.

AIM 1: Participants undergo measurement of height/weight and vital signs (blood pressure, temperature, heart and breathing rate), complete lung function testing (spirometry), undergo an exercise test (cardiopulmonary exercise testing [CPET]), and undergo collection of blood samples on study. Participants may also undergo dual X-ray absorptiometry (DEXA) scan on study.

AIM 2: CLL patients complete aerobic based training program on study. Patients then complete all Aim 1 activities again after completion of aerobic based training program.

AIMS 3-4: Indolent NHL patients undergo measurement of height/weight and vital signs (blood pressure, temperature, heart and breathing rate), complete lung function testing (spirometry), undergo an exercise test (CPET), and undergo collection of blood samples on study. Participants may also undergo DEXA scan on study. Patients undergo muscular strength and functional endurance measurements of hand grip strength, upper body power via weighted chest pass, and leg strength with the timed chair stand test and 6-minute walk test (6MWT). Patients are then randomized to 1 of 2 arms.

ARM I: Patients receive usual care on study.

ARM II: Patients complete aerobic based training program on study. Patients then complete all baseline activities again after completion of aerobic based training program.

AIM 5: All patients from Aims 3-4 will be invited to repeat Aims 3-4 baseline activities.

After completion of study intervention, patients are followed up every 6 months (Aims 2-4) or annually (Aim 5) for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Between the ages of 18-80
* Histologically confirmed diagnosis of indolent non-Hodgkin lymphoma (NHL) will be required to participate in Aim 2 (CLL/SLL only), aim 3 and 4 (indolent NHL) and aim 5 (indolent NHL) of this study

Exclusion Criteria:

* Healthy subjects participating in Aim 1 will be excluded if they have known cardiovascular or pulmonary disease (e.g. heart disease, coronary artery disease, chronic obstructive pulmonary disease [COPD], asthma, etc.) an orthopedic or musculoskeletal limitation which would limit ability to exercise or are a current or former smoker
* Indolent NHL individuals receiving treatment must have least 8 weeks of planned treatment remaining and those who have already received treatment must be at least 6 months post and have no planned treatments during the 12-week intervention period to be eligible. Individuals that are participating prior to receiving treatment must not have any scheduled treatments during their participation. Individuals will be excluded if they have uncontrolled hypertension, cardiac illness, or are not approved by their oncologist to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2028-03-13 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Assess circulating immune cell abundance and function pre-intervention | Baseline
  A standardized questionnaire will be administered to assess levels of past and current physical activity. Baseline measurement of pulmonary function (PFT) will be collected and possibly a body composition scan via dual x-ray absorptiometry (DEXA). While subjects perform cardiopulmonary exercise testing (CPET), cardiopulmonary vitals will be assessed and monitored throughout exercise and in recovery. A 40 mL venous blood sample will be drawn at baseline and post exercise (80 mL total), along with finger prick measures of blood lactate at rest and early recovery. Blood samples will be evaluated to determine how circulating immune cell abundance and function (via cell counts & cytokine profile) of chronic lymphocytic leukemia (CLL) patients respond to acute (single bout) maximal exercise and how this differs from the response observed in group of age-matched controls by monitoring cardiopulmonary parameters and mobilization of immune cell phenotypes.
Assess circulating immune cell mobilization and function post-intervention | Up to 12 weeks
  Each subject will participate in a 12-weeks exercise program (3 times per week) at a moderate to high exercise intensity level based upon the results of their cardiopulmonary exercise testing (CPET)]. Upon completion of the program, subjects will return to the laboratory for post testing using the same techniques as used during the baseline. Venous blood samples drawn at rest after the program will be used to determine how circulating immune cell mobilization and function (cell counts and cytokine profile) of CLL patients respond to intervention. Usual descriptive statistics will be performed - means, standard deviations, and ranges. Comparisons within a group over time or pre/post will be performed using paired t-tests, while comparisons between groups will be performed using unpaired t-tests or where necessary using ANOVA. Comparisons will be made based on absolute values as well as changes during a test.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Gustafson, PhD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials